CLINICAL TRIAL: NCT05430815
Title: Minding the Gap: Improving Women's Health Through Coordinated Postpartum Planning
Brief Title: Improving Women's Health Through Coordinated Postpartum Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Anne Lang Dunlop, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00001427; 1R01MD016031 (NIH)
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Maternal Death; Maternal Morbidity
Keywords: Maternal mortality; Severe maternal morbidity; Postpartum care
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Information on all outpatient visits occurring between delivery discharge and 12 weeks postpartum will be abstracted and blinded for review. Two independent physicians will review the blinded information and determine whether the visit meets the criteria for a comprehensive postpartum visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Postpartum Care System (Experimental): Women with a documented diagnosis of chronic diabetes, chronic hypertension, gestational diabetes, hypertensive disorder of pregnancy (gestational hypertension or preeclampsia), or pre-pregnancy obesity who are randomized to receive enhanced postpartum care.
  Interventions: Behavioral: Enhanced Postpartum Care System
- Standard of Care (No Intervention): Women with a documented diagnosis of chronic diabetes, chronic hypertension, gestational diabetes, or hypertensive disorder of pregnancy (gestational hypertension or preeclampsia), or pre-pregnancy obesity who are randomized to receive standard postpartum care.

INTERVENTIONS:
Behavioral: Enhanced Postpartum Care System — The intervention consists of a comprehensive postpartum care system that integrates American College of Obstetrician and Gynecologist's (ACOG) postpartum care guidelines together with American College of Cardiology and American Heart Association (ACC/AHA) guidelines for the prevention of cardiovascular disease in women, as well as patient preferences for care coordination and communication. The system consists of: 1) a tailored postpartum care plan that is collaboratively developed with patient and provider input and addresses both social and medical needs; 2) an electronic medical record (EMR) based tool for documenting the plan and monitoring postpartum care; and 3) a postpartum follow-up phone call at 1 week postpartum.
  Arms: Enhanced Postpartum Care System

SUMMARY:
The purpose of the study is to design, implement, and evaluate a holistic postpartum women's health care system for women who have cardiovascular risk factors for severe maternal morbidity (SMM) including chronic hypertension, chronic diabetes, gestational diabetes, pre-pregnancy obesity, or a hypertensive disorder of pregnancy (HDP) which includes gestational hypertension or preeclampsia. The researchers will use a sequential mixed methods design. First, the researchers will conduct in-depth interviews with women who have given birth in the prior year to characterize barriers and facilitators to accessing postpartum care. The information from these interviews will be used to inform the design of a postpartum care system. Next, the researchers will conduct a pragmatic randomized trial to test the effectiveness of the system on postpartum care engagement versus standard of care.

DETAILED DESCRIPTION:
The US maternal mortality ratio is the highest among developed nations at 26.4 maternal deaths per 100,000 livebirths. Among the states, Georgia has the second highest maternal mortality (66.3 per 100,000), with a 60% higher rate for black vs white women (95.6 vs 59.7 per 100,000). Nearly 100 times more common than maternal mortality is severe maternal morbidity (SMM), defined as unexpected outcomes of labor and delivery that result in short- and long-term deleterious health consequences. Maternal mortality and SMM are highest among women who are black, publicly insured or uninsured, and deliver in safety-net hospitals. In Georgia, 66% of maternal deaths occur to women insured by Medicaid at delivery and the majority of deaths and SMM occur postpartum, a time during which healthcare visits are poorly attended and oftentimes inaccessible. The Georgia Maternal Mortality Review Committee concluded that two-thirds of maternal deaths are preventable, with chronic health conditions, obesity, delays in accessing and fragmentation of care as key contributors. As solutions, it recommends improved prenatal and postpartum follow-up and case management, control of chronic health conditions, and extension of Medicaid coverage beyond 60 days postpartum.

While the postpartum period represents a crucial window of opportunity for promoting women's current and future health, up to 40% of US women do not attend postpartum visits due to structural barriers (e.g., lack of insurance, transportation or childcare) social barriers (e.g., medical mistrust and poor patient-provider relationships) or low perceived utility of postpartum care. Moreover, the lowest rates of postpartum care utilization are concentrated among women with the highest rates of pregnancy complications and chronic conditions (e.g., women who are uninsured or Medicaid-insured, low-income, and non-Hispanic black). Timely and adequate use of postpartum care is especially important for women with diabetes or hypertensive disease as these conditions are associated with increased risk for postpartum morbidity and mortality and cardiovascular disease later in life.

The researchers of this study plan to conduct an intervention study to assess the effect of a woman-centered, comprehensive postpartum care system on postpartum visit attendance and follow-up care among medically underserved women with chronic diabetes, chronic hypertension, gestational diabetes, pre-pregnancy obesity or hypertensive disorder of pregnancy (HDP). Because implementing and sustaining a comprehensive postpartum care system in a health disparities population requires a thorough understanding of patient preferences regarding the structural and process elements of care, methods of provider-patient communication, and strategies for addressing social and contextual barriers to care the researchers will use in-depth interviews to inform the intervention design and then assess health outcomes and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women between 20-34 weeks of gestation
* have received 1 or more prenatal care visits at Grady Memorial Hospital in Atlanta, Georgia (GA)
* intend to deliver at Grady Memorial Hospital
* speak English or Spanish
* have a diagnosis of chronic diabetes, chronic hypertension, gestational diabetes, pre-pregnancy obesity (body mass index [BMI] of 30 or greater), and/or a hypertensive disorder of pregnancy (gestational hypertension or preeclampsia) documented in the electronic medical record (EMR)

Exclusion Criteria:

* adults unable to consent, infants, and prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dunlop, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The final fully deidentified dataset that will be made available for sharing will include sociodemographic, health behavioral, and health care utilization data from both questionnaire and medical record abstraction, to include race/ethnicity, age, insurance type, visits to health care provider/clinic/or hospital within one year postpartum, including any diagnoses, medical testing and/or laboratory screenings (and results of those tests), prescribed medications and adherence to prescribed medications, as well as data related to any subsequently conceived pregnancy.
Supporting Information: Study Protocol
Time Frame: Data will become available one year after study completion (starting May 1, 2025) and will be made available for 5 years (through April 30, 2030).
Access Criteria: The researchers will make the data and associated documentation available to users under a data-sharing agreement. Outside researchers must submit a Data Analysis Request Form, which requires elucidation of the specific data requested along with a statement that the investigator must provide: 1) a commitment to using the data only for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The Data Analysis Request Form will be made web-accessible with directions to submit the request for review. Outside investigators must have satisfactorily completed a Data Use and Confidentiality Agreement, before the anonymized data is released.

REFERENCES:
- [Derived] Stanhope KK, Stallworth T, Forrest AD, Vuncannon D, Juarez G, Boulet SL, Geary F, Dunlop AL, Blake SC, Green VL, Jamieson DJ. Planning for the forgotten fourth trimester of pregnancy: A parallel group randomized control trial to test a postpartum planning intervention vs. standard prenatal care. Contemp Clin Trials. 2024 Aug;143:107586. doi: 10.1016/j.cct.2024.107586. Epub 2024 Jun 3. PMID 38838985

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Postpartum Care System: Women with a documented diagnosis of chronic diabetes, chronic hypertension, gestational diabetes, hypertensive disorder of pregnancy (gestational hypertension or preeclampsia), or pre-pregnancy obesity randomized to receive enhanced postpartum care.
  Enhanced Postpartum Care System consists of a comprehensive postpartum care system that integrates American College of Obstetrician and Gynecologist's (ACOG) postpartum care guidelines together with American College of Cardiology and American Heart Association (ACC/AHA) guidelines for the prevention of cardiovascular disease in women, as well as patient preferences for care coordination and communication. The system consists of: 1) a tailored postpartum care plan that is collaboratively developed with patient and provider input and addresses both social and medical needs; 2) an electronic medical record (EMR) based tool for documenting the plan and monitoring postpartum care; and 3) a postpartum follow-up phone call at 1 week postpartum.
- Standard of Care: Women with a documented diagnosis of chronic diabetes, chronic hypertension, gestational diabetes, or hypertensive disorder of pregnancy (gestational hypertension or preeclampsia), or pre-pregnancy obesity randomized to receive standard postpartum care.
Period: Overall Study
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Started | 159 | 161
Completed Assessment at 12 Weeks Post-delivery | 141 | 141
Completed (Completed assessment at 14 months post-delivery) | 124 | 117
Not Completed | 35 | 44

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Postpartum Care System: Women with a documented diagnosis of chronic diabetes, chronic hypertension, gestational diabetes, hypertensive disorder of pregnancy (gestational hypertension or preeclampsia), or pre-pregnancy obesity randomized to receive enhanced postpartum care.
- Total: Total of all reporting groups
Arm/Group | Enhanced Postpartum Care System | Standard of Care | Total
Number analyzed (Participants) | 159 | 161 | 320
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 42 | 37 | 79
  25-34 | 81 | 78 | 159
  35-45 | 36 | 46 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 161 | 320
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 23 | 46
  Not Hispanic or Latino | 136 | 138 | 274
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 133 | 131 | 264
  White | 3 | 5 | 8
  More than one race | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 159 | 161 | 320
Type of health insurance at delivery [Count of Participants; unit: Participants]
  Medicaid/Medicare | 119 | 132 | 251
  Private insurance | 35 | 27 | 62
  Self-pay | 1 | 1 | 2
  Unknown | 4 | 1 | 5
Gestational age at study enrollment [Count of Participants; unit: Participants]
  20-27 weeks | 98 | 97 | 195
  28-34 weeks | 61 | 64 | 125
Documented diagnoses [Count of Participants; unit: Participants]
  Chronic hypertension | 70 | 70 | 140
  Diabetes mellitus | 18 | 21 | 39
  Pre-pregnancy obesity | 79 | 70 | 149
  Gestational diabetes | 18 | 24 | 42
  Hypertensive disorders of pregnancy | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending a Comprehensive Postpartum Visit
Description: The postpartum visit occurs between 4 and 12 weeks after delivery and meets specific, defined as a preventive care visit with an obstetric care provider (e.g., obstetrician-gynecologist, certified nurse midwife, or primary care provider with additional training relevant to postpartum care) that included an assessment of assessing multiple aspects of physical and mental health. Comprehensive postpartum visit attendance was identified using data from medical records using a standardized abstraction form.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants | 84 | 89

2. Secondary Outcome: Number of Participants Attending Any Postpartum Visit
Description: Any type of outpatient postpartum visit between 4 and 12 weeks after delivery other than visits to urgent care and/or emergency departments. Postpartum visit attendance was identified using data from medical records using a standardized abstraction form.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants | 109 | 116

3. Secondary Outcome: Number of Participants for Whom Postpartum Diabetes Screening Was Ordered
Description: Any health care provider order of a postpartum screening for diabetes through laboratory testing was identified using data from medical records.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants
  Postpartum diabetes screening ordered | 18 | 26
  Postpartum diabetes screening not ordered | 141 | 135

4. Secondary Outcome: Number of Participants for Whom Postpartum Diabetes Screening Was Performed
Description: Any completed postpartum screening for diabetes through laboratory testing was identified using data from medical records.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants
  Postpartum diabetes screening completed | 9 | 14
  Postpartum diabetes screening not completed | 150 | 147

5. Secondary Outcome: Number of Participants With Diabetes for Whom Postpartum Diabetes Screening Was Ordered
Description: Any health care provider order of a postpartum screening for diabetes through laboratory testing was identified using data from medical records, among enrolled participants diagnosed with gestational diabetes or diabetes mellitus.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants diagnosed with gestational diabetes or diabetes mellitus.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 36 | 45
Participants
  Postpartum diabetes screening ordered | 14 | 19
  Postpartum diabetes screening not ordered | 22 | 26

6. Secondary Outcome: Number of Participants With Diabetes for Whom Postpartum Screening Was Performed
Description: Any completed postpartum screening for diabetes through laboratory testing was identified using data from medical records, among enrolled participants diagnosed with gestational diabetes or diabetes mellitus.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants diagnosed with gestational diabetes or diabetes mellitus.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 36 | 45
Participants
  Postpartum diabetes screening completed | 8 | 11
  Postpartum diabetes screening not completed | 28 | 34

7. Secondary Outcome: Number of Participants Receiving Postpartum Hypertension Screening
Description: Receipt of early postpartum screening (within 0 to 3 weeks of delivery) for hypertension through blood pressure medications identified using data from medical records.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants | 80 | 81

8. Secondary Outcome: Number of Participants With Hypertension Receiving Postpartum Hypertension Screening
Description: Receipt of early postpartum screening (within 0 to 3 weeks of delivery) for hypertension through blood pressure medications identified using data from medical records, among enrolled participants diagnosed with hypertensive disorders of pregnancy or chronic hypertension.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants diagnosed with hypertensive disorders of pregnancy or chronic hypertension.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 75 | 78
Participants | 45 | 48

9. Secondary Outcome: Number of Participants Using Contraception 12 Weeks After Delivery
Description: The number of participants using contraception is evaluated via patient self-report survey.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants who completed the assessment at 12 weeks post-delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 141 | 141
Participants | 119 | 117

10. Secondary Outcome: Number of Participants Using Contraception 14 Months After Delivery
Description: The number of participants using contraception is evaluated via patient self-report survey.
Time Frame: 14 months after delivery
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants Using Medication 12 Weeks After Delivery
Description: The number of participants using prescription medication for chronic conditions is evaluated via medical record abstraction.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants | 21 | 29

12. Secondary Outcome: Number of Participants Using Medication 14 Months After Delivery
Description: The number of participants using prescription medication for chronic conditions will be evaluated via medical record abstraction.
Time Frame: 14 months after delivery
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants With Ongoing Pregnancy Complications at 12 Weeks After Delivery
Description: The number of participants with diagnoses of severe maternal morbidity since the birth of their baby, identified from medical records using International Classification of Diseases diagnosis and any procedure codes from readmissions following the delivery.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants | 2 | 3

14. Secondary Outcome: Number of Participants With Ongoing Pregnancy Complications at 14 Months After Delivery
Description: as for outcome 13
Time Frame: 14 months after delivery
Reporting Status: Not Posted

15. Secondary Outcome: Number of Participants Readmitted to the Hospital at 12 Weeks After Delivery
Description: The number of participants with any medical complication(s) resulting in hospital readmission since the birth of their baby.
Time Frame: 12 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 159 | 161
Participants | 6 | 9

16. Secondary Outcome: Number of Participants Readmitted to the Hospital at 14 Months After Delivery
Description: as for outcome 15
Time Frame: 14 months after delivery
Reporting Status: Not Posted

17. Secondary Outcome: Perceived Risk of Severe Maternal Morbidity (SMM)
Description: Future severe maternal morbidity risk perception is assessed with a single question asking participants if they think they are at higher or lower risk of having a serious pregnancy complication during a future pregnancy compared to other women of the same age. Responses are given on a 3-point scale where 1 = low risk and 3 = high risk.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants who completed the assessment at 12 weeks post-delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 141 | 141
Participants
  Perceived risk value - low risk | 35 | 34
  Perceived risk value - average or high risk | 66 | 76
  Don't know/refused to answer/missing response | 40 | 31

18. Secondary Outcome: Perceived Risk of Cardiovascular Disease at 12 Weeks After Delivery
Description: Future cardiovascular disease risk perception is assessed with a single question asking participants if they think they are at higher or lower risk of having a heart attack or stroke compared to other women of the same age. Responses are given on a 3-point scale where 1 = low risk and 3 = high risk.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants who completed the assessment at 12 weeks post-delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 141 | 141
Participants
  Low risk | 55 | 58
  Average or high risk | 26 | 31
  Don't know/refused to answer/missing response | 60 | 52

19. Secondary Outcome: Perceived Risk of Cardiovascular Disease at 14 Month After Delivery
Description: as for outcome 18
Time Frame: 14 months after delivery
Reporting Status: Not Posted

20. Secondary Outcome: Number of Participants Using Primary Care
Description: The number of participants planning to attend, or have already attended, a visit with a primary care provider will be evaluated via medical record abstraction 14 months after delivery.
Time Frame: 14 months after delivery
Reporting Status: Not Posted

21. Secondary Outcome: Number of Participants Using Specialty Care
Description: The number of participants planning to attend, or having already attended, a visit with a specialty health care will be evaluated via medical record abstraction 14 months after delivery.
Time Frame: 14 months after delivery
Reporting Status: Not Posted

22. Secondary Outcome: Number of Participants With Depression Per Edinburgh Postnatal Depression Scale (EPDS) Score at 12 Weeks After Delivery
Description: Depressive symptoms are assessed with the Edinburgh Postnatal Depression Scale (EPDS). The EPDS includes 10-items asking participants about symptoms of depression that they have experienced in the past 7 days. Responses are given on a 4-point scale where 0 corresponds with the least amount of symptoms and 3 corresponds with the highest amount of symptoms. Total scores range from 0 to 30 with higher scores indicating increased symptoms of depression. Scores of 13 or greater indicate that the respondent is likely suffering from depression.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants who completed the assessment at 12 weeks post-delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 141 | 141
Participants
  EPDS score of 13 or higher | 37 | 26
  EPDS score of less than 13 | 88 | 92
  Refused to answer/missing response | 16 | 23

23. Secondary Outcome: Number of Participants With Depression Per Edinburgh Postnatal Depression Scale (EPDS) Score at 14 Months After Delivery
Description: as for outcome 22
Time Frame: 14 months after delivery
Reporting Status: Not Posted

24. Secondary Outcome: Satisfaction With Postpartum Care
Description: Satisfaction with the postpartum checkup is assessed by asking those participants who reported completing a postpartum visit if they were satisfied with the wait time, amount of time with healthcare providers, advice given, and respect shown to each individual as a person. Responses are given as "yes" or "no". The count of participants reporting satisfaction with each separate item is assessed.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants who reported completing a postpartum visit. Some participants did not respond to every survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 95 | 90
Participants
  Satisfied with wait time: number analyzed (Participants) | 93 | 89
  Satisfied with wait time | 88 | 81
  Satisfied with amount of time with healthcare providers: number analyzed (Participants) | 93 | 89
  Satisfied with amount of time with healthcare providers | 90 | 79
  Satisfied with advice given: number analyzed (Participants) | 94 | 89
  Satisfied with advice given | 91 | 82
  Satisfied with respect shown to each individual as a person | 93 | 87

25. Secondary Outcome: Satisfaction With Provider at Postpartum Care Visit
Description: Satisfaction with the healthcare provider at the postpartum care visit is assessed with 4 items. Responses are given on a 5-point scale where 1 = poor and 5 = excellent. Each item is scored separately and higher scores indicate greater satisfaction with the healthcare provider.
Time Frame: 12 weeks after delivery
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 95 | 90
units on a scale
  Respected me as a person | 4.7 (0.6) | 4.7 (0.5)
  Letting me say what mattered to me about my health: number analyzed (Participants) | 94 | 89
  Letting me say what mattered to me about my health | 4.7 (0.6) | 4.6 (0.8)
  Taking my preferences seriously: number analyzed (Participants) | 95 | 88
  Taking my preferences seriously | 4.7 (0.7) | 4.6 (0.8)
  Giving me enough information to make the best decisions about my health: number analyzed (Participants) | 95 | 88
  Giving me enough information to make the best decisions about my health | 4.7 (0.6) | 4.6 (0.9)

26. Secondary Outcome: Number of Participants in Self-rated Categories of Postpartum Health at 12 Weeks After Delivery
Description: Participants are asked to self-rate their perception of their physical health and mental health since delivery as "excellent", "very good", "good", "fair", "declined" or "poor". The number of participants endorsing each category of health is presented.
Time Frame: 12 weeks after delivery
Population: This analysis includes participants who completed the assessment at 12 weeks post-delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Postpartum Care System | Standard of Care
Number analyzed (Participants) | 141 | 141
Participants
  Physical Health Since Delivery: Excellent | 47 | 50
  Physical Health Since Delivery: Very Good | 18 | 23
  Physical Health Since Delivery: Good | 43 | 32
  Physical Health Since Delivery: Fair | 23 | 24
  Physical Health Since Delivery: Declined | 1 | 2
  Physical Health Since Delivery: Poor | 5 | 3
  Physical Health Since Delivery: Missing response/refused to answer | 4 | 7
  Mental health since delivery: Excellent | 49 | 53
  Mental health since delivery: Very Good | 21 | 22
  Mental health since delivery: Good | 26 | 29
  Mental health since delivery: Fair | 28 | 24
  Mental health since delivery: Declined | 6 | 3
  Mental health since delivery: Poor | 8 | 9
  Mental health since delivery: Missing response/refused to answer | 3 | 1

27. Secondary Outcome: Number of Participants in Self-rated Categories of Postpartum Health at 14 Months After Delivery
Description: as for outcome 26
Time Frame: 14 months after delivery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of informed consent and continued through the first 12 weeks after delivery, and through the final assessment at 14 months after delivery.
Description: In this study, non-serious adverse events are defined as events graded as moderate or higher that resulted in participants seeking care at an emergency department or urgent care center. Serious Adverse Events (SAEs) were defined as: death, a life-threatening event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, a congenital anomaly or birth defect, or an important medical event based upon appropriate medical judgment.
Arm/Group | Enhanced Postpartum Care System | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/161
Serious Adverse Events (participants affected / at risk) | 6/159 | 9/161
Other Adverse Events (participants affected / at risk) | 39/159 | 27/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enhanced Postpartum Care System (N=159) | Standard of Care (N=161)
Inpatient hospitalization through 12 weeks postpartum for sepsis (Pregnancy, puerperium and perinatal conditions) | 2 | 1 — Severe maternal morbidity event
Inpatient hospitalization through 12 weeks postpartum for preeclampsia (Pregnancy, puerperium and perinatal conditions) | 4 | 2
Inpatient hospitalization through 12 weeks postpartum for eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Severe maternal morbidity event
Inpatient hospitalization through 12 weeks postpartum for cerebral hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Severe maternal morbidity event
Inpatient hospitalization through 12 weeks postpartum for endometriosis (Reproductive system and breast disorders) | 0 | 1
Inpatient hospitalization through 12 weeks postpartum for cholecystitis (Hepatobiliary disorders) | 0 | 1
Inpatient hospitalization through 12 weeks postpartum for small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Inpatient hospitalization through 12 weeks postpartum for colostomy reversal (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enhanced Postpartum Care System (N=159) | Standard of Care (N=161)
Vaginal bleeding (Reproductive system and breast disorders) | 1 | 2
Breastfeeding issues (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Mental health issues (Psychiatric disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Hypertension (Vascular disorders) | 7 | 6
New pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Genitourinary infection (Infections and infestations) | 4 | 0
Wound dehiscence or minor infection (Surgical and medical procedures) | 6 | 5
Acute upper respiratory, skin, or dental infection (Infections and infestations) | 10 | 6
Chronic condition exacerbation (General disorders) | 3 | 2
Acute cholecystitis (Hepatobiliary disorders) | 2 | 0
Family planning (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT05430815/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/15/NCT05430815/ICF_000.pdf